CLINICAL TRIAL: NCT06772441
Title: Prostate-only, Dose-escalated Radiotherapy Plus Concomitant Androgen Deprivation Therapy in Primary Localized, NCCN High Risk and MMAI Classifier Low or Intermediate-risk Prostate Cancer - a Prospective, Single-arm, Phase II Study
Brief Title: Artificial Intelligence Driven Personalisation of Radiotherapy and Concomitant Androgen Deprivation Therapy for Prostate Cancer Patients (the HypoPro Trial)
Acronym: HypoPro
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: German Oncology Center, Cyprus (Other)
Collaborators: Artera (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-PRC-062; 2024-510707-11-00 (EU CTIS Number); U1111-1309-9298 (Other: World Health Organization UTN)
Record Dates: First submitted 2025-01-03; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer
Keywords: artificial intelligence; ADT; radiation therapy; androgen deprivation therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single experimental arm (Experimental): Prostate +/-seminal vesicles base HDR BT with 15 Gy (D90) / 1 fraction followed by SBRT with 25 Gy in 5 Gy / fraction (daily); of the prostate +- seminal vesicles. Concomittant/adjuvant admission of 12 months ADT.
  Interventions: Drug: Androgen deprivation therapy (ADT)

INTERVENTIONS:
Drug: Androgen deprivation therapy (ADT) — * Goserelin: AstraZeneca, 10.8mg injection
  * ADT will be applied for 12 months in total
  * ADT must be given concurrently and adjuvant

SUMMARY:
The aim of this prospective, single-arm phase II study is the individualization of both radiotherapy (RT) and androgen deprivation therapy (ADT) duration for patients with high-risk localized prostate cancer (PCa) according to the National Comprehensive Cancer Network (NCCN) based on multimodal artificial intelligence (MMAI) classification. All patients will receive (i) a dose escalation to the prostate via HDR brachytherapy (boost), (ii) twelve months of ADT and (iii) extremely hypofractionated RT to the prostate (5 fractions).

This way, patients in the HypoPro trial will receive a prostate-only dose escalation and benefit from shortening of the ADT compared with current guideline recommendations.

DETAILED DESCRIPTION:
In Cyprus approximately 800 men are newly diagnosed with PCa every year. Prostate cancer caused 6.1 million disability-adjusted life-years (DALYs) globally in 2016. The socio-economic burden is high since PCa-related life-time costs are approximately 40,000 per patient with early stage disease at initial diagnosis.

This is a prospective, single-center phase II trial. Patient participants will receive treatment for prostate +-seminal vesicles base high-dose-rate brachytherapy (HDR BT) with 15 Gray units (Gy) with minimal dose covering 90% of the prostate (D90) / 1 fraction followed by stereotactic body radiation therapy (SBRT) with 25 Gy in 5 Gy / fraction (daily); of the prostate +- seminal vesicles. Concomittant/adjuvant admission of 12 months ADT.

First: 1 fraction HDR BT including fiducial placement Second: 14 ±2 days gap Third: 5 fractions of SBRT within 5 consecutive weekdays For the HypoPro patients, we expect no significant differences in disease-free survival (DFS) rates compared to the FLAME trial (2) which one arm treated the patients with moderately-hypofractionated RT to the prostate plus dose escalation to the intraprostatic tumor plus 18-24 months of ADT. Secondary endpoints like metastatic free survival, prostate cancer survival and overall survival will depict the oncologic efficacy in this patient cohort. Thus, the results of this study might be used as the basis for a randomized-controlled trial comparing this dose escalated radiotherapy plus shortened ADT duration with the standard of care (no dose escalated RT, ADT for 2-3 years) in this highly selected treatment group: NCCN high-risk, prostate-specific membrane antigen (PSMA) positron emission tomography (PET) cN0/cM0 and MMAI low/intermediate-risk. Considering the epidemiological importance of the PCa, these results could have a significant socio-economic impact. In parallel a translational research program will address the identification of novel biomarkers to predict the treatment outcome.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed adenocarcinoma of the prostate (histological confirmation can be based on tissue taken at any time, but a re-biopsy should be considered if the biopsy is more than 12 months old)
2. Primary PCa (in PSMA-PET imaging and multiparametric magnetic resonance imaging (mpMRI)
3. High-risk according to NCCNv4.2023 criteria (cT3a or Grade group 4-5 or PSA > 20 ng/ml)
4. Signed written informed consent for this study
5. Age >18 years
6. Previously conducted PSMA-PET/CT, mpMRI or PSMA-PET/MR
7. MMAI low-/intermediate-risk
8. ECOG Performance score 0 or 1
9. IPSS Score ≤15
10. Prostate biopsy core with the highest ISUP grade available

Exclusion Criteria:

1. Prior radiotherapy to the prostate or pelvis
2. Prior radical prostatectomy
3. Prior focal therapy approaches to the prostate
4. Evidence of pelvic nodal disease (cN+) in mpMRI and/or PSMA-PET/CT
5. Evidence of distant metastatic disease (cM+) in mpMRI and/or PSMA-PET/CT
6. Time gap between the beginning of any systemic therapy, ADT and conduction of PSMA-PET scans is >2 months
7. Evidence of cT4 disease in mpMRI and/or PSMA-PET/CT
8. PSA >50 ng/ml prior to starting of systemic therapy
9. Expected patient survival <5 years
10. Bilateral hip prostheses or any other implants/hardware that would introduce substantial CT artifacts
11. Contraindication to undergo a MRI scan
12. Contraindication to undergo HDR brachytherapy (brachytherapy not feasible due to large prostate volume, prostate anatomy, tumor in distant seminal vesicles and/or unfit for anaesthesia)
13. Contraindication to Goserelin
14. Prostate surgery (TURP or HOLEP) with a significant tissue cavity or prostate surgery (TURP or HOLEP) within the last 6 months prior to randomization
15. Medical conditions likely to make radiotherapy inadvisable e.g. acute inflammatory bowel disease, hemiplegia or paraplegia
16. Previous malignancy within the last 2 years (except basal cell carcinoma or squamous cell carcinoma of the skin), or if previous malignancy is expected to significantly compromise 5 year survival
17. Any other contraindication to external beam radiotherapy (EBRT) to the pelvis
18. Participation in any other interventional clinical trial within the last 30 days before the start of this trial
19. Simultaneous participation in other interventional trials which could interfere with this trial; simultaneous participation in registry and diagnostic trials is allowed
20. Patient without legal capacity who is unable to understand the nature, significance and consequences of the trial;
21. Known or persistent abuse of medication, drugs or alcohol
22. Patients expected to have severe set up problems (e.g. mental condition)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Males with prostate cancer. Eligibility is based on histologically confirmed adenocarcinoma of the prostate
Enrollment: 30 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival 5 years after treatment | Five years
  Disease recurrence is defined as PSA failure according to Phoenix, new lesions on PSMA PET and/or MRI imaging or the beginning of any salvage therapy.

SECONDARY OUTCOMES:
Time to local or regional failure, after end of RT | Two and five years after RT
  Local or regional recurrences have to be confirmed by PSMA-PET or mpMR imaging. For the diagnosis of local failure, verification via biopsy is warranted
Metastatic free survival (MFS) after end of RT | Two and five years after RT
  MFS is defined as survival time in months from beginning of RT until detection of any new lesion confirmed as metastasis by PSMA-PET/CT or mpMR imaging or death.
Overall survival (OS) | Assessment at 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 and 60 months after RT
  OS will be measured from the last day of RT to the date of death whatever the cause of death is. Patients who are alive are censored at the date of the most recent follow-up examination. The cause of death of each patient dying during the study will be recorded and reported.
Prostate cancer specific survival (PCSS) | Assessment at 1, 3, 6, 9, 12, 18, 24, 30, 36, 42, 48, 54 and 60 months after RT
  PCSS is defined from the last day of RT until death as most reasonable consequence of progressive prostate cancer, judged by the investigator.
Biochemical failure | Two and five years after RT
  Time to biochemical failure after end of RT (phoenix definition)
Quality of Life (QoL) | Assessment at 6, 9, 12, 18, and 24 months after randomization (± 14 days for each visit) and at 30, 36, 42, 48, 54, 60 months after Ultra-hypofractionated RT - UHF (± 1 month)
  Patient-reported outcome measures (PROMs) EPIC-26: the Expanded Prostate Cancer Index-Short form) with score: 0-100
Quality of Life (QoL) | Assessment at 6, 9, 12, 18, and 24 months after randomization (± 14 days for each visit) and at 30, 36, 42, 48, 54, 60 months after Ultra-hypofractionated RT - UHF (± 1 month)
  Patient-reported outcome measures (PROMs) IIEF-5: The International Index of Erectile Function with score: 0-5
Genitourinary (GU) acute toxicities | During, at 1 and 3 months after RT
  Cumulative acute GU toxicities using the RTOG grading system (Radiation Therapy Oncology Group; with grade: 0-5, where 0 implies no toxicity and 5 implies a side effect related to death)
GU acute toxicities | During, at 1 and 3 months after RT
  Cumulative acute GU toxicities using the CTCAE v5.0 criteria (the Common Terminology Criteria for Adverse Events criteria; with grade: 1-5 where 1 means asymptomatic or mild symptoms and 5 means death related to adverse event)
GU chronic toxicities | During, at 1 and 3 months after RT
  Cumulative chronic GU toxicities using the RTOG grading system (Radiation Therapy Oncology Group; with grade: 0-5, where 0 implies no toxicity and 5 implies a side effect related to death)
GU chronic toxicities | during, 1 and 3 months after RT
  Cumulative chronic GU toxicities using the CTCAE v5.0 criteria (the Common Terminology Criteria for Adverse Events criteria; with grade: 1-5 where 1 means asymptomatic or mild symptoms and 5 means death related to adverse event)
Gastrointestinal (GI) acute toxicities | During, 1 and 3 months after RT
  Cumulative acute GI toxicities using the RTOG grading system (Radiation Therapy Oncology Group; with grade: 0-5, where 0 implies no toxicity and 5 implies a side effect related to death)
GI acute toxicities | During, at 1 and 3 months after RT
  Cumulative acute GU toxicities using the CTCAE v5.0 criteria (the Common Terminology Criteria for Adverse Events criteria; with grade: 1-5 where 1 means asymptomatic or mild symptoms and 5 means death related to adverse event)
GI chronic toxicities | Assessment at 6, 9, 12, 18, and 24 months after RT
  Cumulative chronic GU toxicities using the RTOG grading system (Radiation Therapy Oncology Group; with grade: 0-5, where 0 implies no toxicity and 5 implies a side effect related to death)
GI chronic toxicities | Assessment at 6, 9, 12, 18, and 24 months after RT
  Cumulative acute GU toxicities using the CTCAE v5.0 criteria (the Common Terminology Criteria for Adverse Events criteria; with grade: 1-5 where 1 means asymptomatic or mild symptoms and 5 means death related to adverse event)
Testosterone recovery | Assessment at 6, 9, 12, 18 and 24 months after randomization (± 14 days for each visit) and at 30, 36, 42, 48, 54, 60 months after Ultra-hypofractionated RT - UHF (± 1 month)
  Testosterone recovery is to be done through a blood test

CONTACTS AND LOCATIONS:
Locations (1):
- German Oncology Center, Limassol, Cyprus

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gorovets D, Hopkins M, Kollmeier M, Moore A, Goel A, Shasha D, Brennan V, McBride S, Cohen G, Damato AL, Zelefsky MJ. Early outcomes of high-dose-rate brachytherapy combined with ultra-hypofractionated radiation in higher-risk prostate cancer. Brachytherapy. 2021 Nov-Dec;20(6):1099-1106. doi: 10.1016/j.brachy.2021.08.006. Epub 2021 Sep 26. PMID 34588146
- [Background] van As N, Griffin C, Tree A, Patel J, Ostler P, van der Voet H, Loblaw A, Chu W, Ford D, Tolan S, Jain S, Camilleri P, Kancherla K, Frew J, Chan A, Naismith O, Armstrong J, Staffurth J, Martin A, Dayes I, Wells P, Price D, Williamson E, Pugh J, Manning G, Brown S, Burnett S, Hall E. Phase 3 Trial of Stereotactic Body Radiotherapy in Localized Prostate Cancer. N Engl J Med. 2024 Oct 17;391(15):1413-1425. doi: 10.1056/NEJMoa2403365. PMID 39413377
- [Background] Spratt DE, Tang S, Sun Y, Huang HC, Chen E, Mohamad O, Armstrong AJ, Tward JD, Nguyen PL, Lang JM, Zhang J, Mitani A, Simko JP, DeVries S, van der Wal D, Pinckaers H, Monson JM, Campbell HA, Wallace J, Ferguson MJ, Bahary JP, Schaeffer EM, Sandler HM, Tran PT, Rodgers JP, Esteva A, Yamashita R, Feng FY. Artificial Intelligence Predictive Model for Hormone Therapy Use in Prostate Cancer. NEJM Evid. 2023 Aug;2(8):EVIDoa2300023. doi: 10.1056/EVIDoa2300023. Epub 2023 Jun 29. PMID 38320143
- [Background] Esteva A, Feng J, van der Wal D, Huang SC, Simko JP, DeVries S, Chen E, Schaeffer EM, Morgan TM, Sun Y, Ghorbani A, Naik N, Nathawani D, Socher R, Michalski JM, Roach M 3rd, Pisansky TM, Monson JM, Naz F, Wallace J, Ferguson MJ, Bahary JP, Zou J, Lungren M, Yeung S, Ross AE; NRG Prostate Cancer AI Consortium; Sandler HM, Tran PT, Spratt DE, Pugh S, Feng FY, Mohamad O. Author Correction: Prostate cancer therapy personalization via multi-modal deep learning on randomized phase III clinical trials. NPJ Digit Med. 2023 Feb 22;6(1):27. doi: 10.1038/s41746-023-00769-z. No abstract available. PMID 36813827
- [Background] Kerkmeijer LGW, Groen VH, Pos FJ, Haustermans K, Monninkhof EM, Smeenk RJ, Kunze-Busch M, de Boer JCJ, van der Voort van Zijp J, van Vulpen M, Draulans C, van den Bergh L, Isebaert S, van der Heide UA. Focal Boost to the Intraprostatic Tumor in External Beam Radiotherapy for Patients With Localized Prostate Cancer: Results From the FLAME Randomized Phase III Trial. J Clin Oncol. 2021 Mar 1;39(7):787-796. doi: 10.1200/JCO.20.02873. Epub 2021 Jan 20. PMID 33471548